CLINICAL TRIAL: NCT06319911
Title: AETOS Shoulder System Post Market Clinical Investigation
Brief Title: AETOS Shoulder System
Status: Recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AETOS 2022.04
Record Dates: First submitted 2024-02-28; First posted 2024-03-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Osteoarthritis; Shoulder Arthritis
Keywords: Shoulder; arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Primary Anatomic: Those subjects who have the AETOS implanted in the Primary Anatomic configuration
  Interventions: Device: AETOS
- Primary reverse: Those subjects who have AETOS implanted in the Reverse configuration
  Interventions: Device: AETOS

INTERVENTIONS:
Device: AETOS — The AETOS Shoulder System will be implanted into the right or left shoulder in the anatomic or reverse configuration

SUMMARY:
The goal of this study is to confirm the safety and performance of the AETOS Shoulder System for USA adoption. This is a prospective, open, adaptive, non-comparative, multi-centre investigation enrolling a maximum of 220 subjects in 2 cohorts (anatomic and reverse) at up to 15 sites. No intra-study comparator group will be included, and there will be no randomization

DETAILED DESCRIPTION:
This study will confirm the safety and performance of the AETOS Shoulder System in anatomic and reverse TSA. Revisions will not be enrolled into this study.

The AETOS Shoulder System is manufactured by Smith & Nephew, Inc., 1450 Brooks Road Memphis, Tennessee 38116 USA, and has been 510k Cleared as of 07Jun2023; therefore, it is considered a post-market product and will be procured through normal commercial channels in the USA. The humeral stem is designed to be used for both Total Shoulder Arthroplasty (TSA) and reverse shoulder arthroplasty procedures. The humeral stems are designed with fins and a porous plasma coating to provide fixation within the proximal humeral metaphysis.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be included in the study:

1. Patient is at least 18 years of age at the time of consent and skeletally mature.
2. Patient is undergoing a primary elective anatomic or reverse shoulder replacement surgery for one of the following indications:

   * Rheumatoid arthritis, and/or
   * Traumatic arthritis (Post Traumatic arthritis), and/or
   * Non-inflammatory degenerative joint disease, and/or
   * Correction of functional deformity.
3. Patient is willing and able to accommodate all study-related procedures and visits detailed in the protocol & cooperate in the standard of care post-operative therapy.
4. Patient is geographically stable and willing to return to the study site for all follow-up visits.
5. Patient has been adequately informed of risks and requirements of the study and is willing and able to provide informed consent for participation.

   -

Exclusion Criteria:

Patients who meet any of the following criteria will not qualify for participation in the trial:

1. Patient has a contraindication to AETOS.
2. Patient is undergoing a revision shoulder replacement surgery including total or partial arthroplasty.
3. Patient is indicated for a Hemiarthroplasty.
4. Patient has traumatic injury or a fracture.
5. Patient has uncontrolled diabetes with a hemoglobin A1C of 7.5 or greater.
6. Patient has comorbidities/conditions that preclude proper healing/fixation of the implant.
7. Patient has poor quality or insufficient bone stock to support the implant.
8. Patient has poor bone quality where there could be considerable migration of the implant and/or a chance of fracture.
9. Patient has rapid joint destruction, marked bone loss or bone resorption (e.g., severe osteoporosis).
10. Patient has osteomalacia.
11. Patient has muscular, neurologic, or vascular deficiencies that may compromise the outcome of the shoulder replacement surgery.
12. Patient has a known sensitivity, allergic reaction, and/or known allergies to one or more of the implanted materials.
13. Patient has a distant foci of infection which may spread to the implant site, active local or systemic infection, sepsis, or osteomyelitis.
14. Patient has an elevation of sedimentation rate, elevation of WBC count, or marked shift in WBC differential count unexplained by other disease.
15. If reverse shoulder arthroplasty, patient has a non-functional deltoid or external rotator muscles.
16. If reverse shoulder arthroplasty, patient has a significant injury to the upper brachial plexus.
17. If reverse shoulder arthroplasty, patient has paralysis of the axillary nerve.
18. Patient is uncooperative, has a neurologic disorder and is not capable of following directions, or is a vulnerable subject per ISO 14155 (i.e., individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response).
19. Patient is pregnant or plans to become pregnant during the follow-up period.
20. Patient has a Body Mass Index (BMI) of >35kg/m2 or a BMI that may compromise the outcome of the shoulder replacement surgery.
21. Patient has anticipated activities which would impose high stresses on the implant and its fixation or has a high likelihood of a fall.
22. Patient is a known smoker, vaper, alcohol abuser, or drug abuser within 180 days of consent.
23. Patient has participated previously in this clinical trial and was withdrawn.
24. Patient is participating in another device or drug trial or observational competitive study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females who are at least 18 years of age at the time of consent, are skeletally mature, and are indicated for primary anatomic or primary reverse will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 2 years
  Implant survivorship at 2 years post operatively defined as absence of device removal or revision of any component

SECONDARY OUTCOMES:
Implant Survivorship at 6 months, 1 year, 3.5 years and 5 years | 6 months, 1 year, 3.5 years, and 5 years
  Implant Survivorship at 6 months, 1 year, 3.5 years, and 5 years defined as absence of device removal or revision of any component
Radiographic Assessment - Glenoid Migration/Subsidence | Day 0, 1 year, 2 years, and 5 years
  Glenoid Component Migration / Subsidence collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Absent: No evidence of glenoid component displacement ≥ 5 mm relative to the native bone stock.
  1. Present: Presence of glenoid component displacement ≥ 5 mm relative to the native bone stock.
Radiographic Assessment - Glenoid Radiolucency | Day 0, 1 year, 2 years, and 5 years
  Glenoid Component Radiolucency - antero-posterior (AP) collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Absent: No evidence of radiolucency > 2 mm in width along the bone-implant / bone-cement interface in any zone.
  1. Present: Presence of radiolucency > 2 mm in width along the bone-implant / bone-cement interface in one or more zones.
Radiographic Assessment - Humeral Radiolucency | Day 0, 1 year, 2 years, and 5 years
  Humeral Component Radiolucency - AP collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Absent: No evidence of radiolucency > 2 mm in width along the bone-implant interface in any zone.
  1. Present: Presence of radiolucency > 2 mm in width along the bone-implant interface in one or more zones.
Radiographic Assessment - Humeral Migration/Subsidence | Day 0, 1 year, 2 years, and 5 years
  Humeral Component Migration / Subsidence collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Absent: No evidence of a change in position of the humeral component relative to the native bone stock ≥ 5 mm.
  1. Present: Presence of a change in position of the humeral component relative to the native bone stock ≥ 5 mm
Radiographic Assessment - Humeral Head Centeredness | Day 0, 1 year, 2 years, and 5 years
  Humeral Head Centeredness collected post-surgery at day 0, 1 year, 2 years, and 5 years will be calculated using the method described by Iannotti and Norris from the axillary view
Radiographic Assessment - Bone Remodeling | Day 0, 1 year, 2 years, and 5 years
  Bone Remodeling of the humerus collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions by Schnetzke et al.:
  0. Absent: No evidence of humerus bone remodeling.
  1. Present: Presence of one or more features of humerus bone remodeling.
  * 1. Condensation Lines: Presence of condensation lines around the tip of the stem.
  * 2. Cortical Thinning: Presence of cortical thinning and osteopenia.
  * 3. Spot Welds: Presence of spot welds.
  * 4. Other: Other feature not listed above.
Radiographic Assessment - Glenohumeral Subluxation | Day 0, 1 year, 2 years, and 5 years
  Glenohumeral Subluxation collected post-surgery at day 0, 1 year, 2 years, and 5 years will be will be derived from the Humeral Head Centeredness assessment using the following definitions, from Iannotti and Norris et al.:
  0. Absent: Humeral Head Centeredness is ≤25%.
  1. Present: Humeral Head Centeredness is >25%.
Radiographic Assessment - Device Condition: Anatomic | Day 0, 1 year, 2 years, and 5 years
  Device Condition - Anatomic collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Intact: No evidence of fracture, breakage, loosening, disassembly or migration of any of the components of the anatomic AETOS TSA.
  1. Not Intact: Presence of fracture, breakage, loosening, disassembly or migration of one or more of the components of the anatomic AETOS TSA:
  * 1. Humeral Stem.
  * 2. Humeral Head.
  * 3. Glenoid.
  * 4. Post Extension.
Radiographic Assessment - Device Condition: Reverse | Day 0, 1 year, 2 years, and 5 years
  Device Condition - Reverse collected post-surgery at day 0, 1 year, 2 years, and 5 years will be graded in accordance with the following definitions:
  0. Intact: No evidence of fracture, breakage, loosening, disassembly or migration of any of the components of the reverse AETOS TSA.
  1. Not Intact: Presence of fracture, breakage, loosening, disassembly or migration of one or more of the components of the reverse AETOS TSA:
  * 1. Humeral Stem.
  * 2. Reverse Liner.
  * 3. Glenosphere.
  * 4. Metal Glenoid.
  * 5. Peripheral Screws.
  * 6. Central Screw.
  * 7. Humeral Spacer.
  * 8. Post Extension.
American Shoulder and Elbow Score (ASES) | 6 months, 1 year, 2 years, and 5 years
  The ASES instrument is composed of 2 sections containing participant self-reported and clinician assessments. The ASES score is a 0 to 100-point rating with a higher score indicating improvement in pain and function.
Constant Murley Score | 6 months, 1 year, 2 years, and 5 years
  Constant-Murley Shoulder (CMS) scale assesses four aspects related to shoulder pathology; two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65, resulting in a possible maximum total score of 100 points (best function). Pain and ADL are answered by the subject; ROM and strength require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist.
Simple Shoulder Test (SST) | 6 months, 1 year, 2 years, and 5 years
  Series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answer to these questions provides a standardized way of recording the function of a shoulder before and after treatment.
Single Assessment Numeric Evaluation (SANE) | 6 months, 1 year, 2 years, and 5 years
  The SANE is a simple, single-question, patient-based shoulder function assessment tool: ''How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?''

CONTACTS AND LOCATIONS:
Overall Officials: Kolja Boese, Study Director — Smith & Nephew, Inc.
Locations (5):
- United States (5):
  - California Pacific Orthopedics, San Francisco, California
  - Western Orthopaedics, Denver, Colorado
  - Hughston Foundation, Columbus, Georgia
  - Center for Orthopedics and Neurosurgical Care, Bend, Oregon
  - Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No